CLINICAL TRIAL: NCT01256359
Title: A Double Blind Randomised Phase 2 Trial of Docetaxel With or Without AZD6244 in wt BRAF Advanced Melanoma
Brief Title: Docetaxel With or Without AZD6244 in Melanoma
Acronym: DOC-MEK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OCTO_015
Record Dates: First submitted 2010-11-17; First posted 2010-12-08 (Estimated); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Docetaxel; AZD 6244

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel and AZD6244 (Experimental): Docetaxel with AZD6244
  Interventions: Drug: Docetaxel and AZD6244
- Docetaxel and Placebo (Experimental): Docetaxel without AZD6244
  Interventions: Drug: Docetaxel and placebo

INTERVENTIONS:
Drug: Docetaxel and AZD6244 — Docetaxel 75mg/m2 IV and AZD6244 75mg bd daily. Docetaxel will be administered every 3 weeks for a maximum 6 cycles, but AZD6244 may be continued beyond this, until disease progression.
  Other Names: Taxotere
  Arms: Docetaxel and AZD6244
Drug: Docetaxel and placebo — Docetaxel 75mg/m2 IV and placebo given bd. Docetaxel will be administered every 3 weeks for a maximum 6 cycles, but placebo may be continued beyond this, until disease progression.
  Other Names: Taxotere
  Arms: Docetaxel and Placebo

SUMMARY:
This is a randomised, double-blind placebo controlled phase 2 trial. Patient will be randomly assigned 1:1 between 2 treatment arms. They will receive either docetaxel 75mg/m2 IV and placebo given bd, or AZD6244 75mg bd daily with docetaxel 75mg/m2 IV. Docetaxel will be administered every 3 weeks for a maximum 6 cycles, but AZD6244/placebo may be continued beyond this, until disease progression. The objective is to assess whether the combination of AZD6244 with docetaxel is worthy of evaluation in a definitive randomised study, with the null hypothesis being that the combination has activity similar to that of docetaxel alone in this population. After consent has been obtained mutational analysis of tumour BRAF will be performed on archival tumour tissue, where this information is not already known, to assess eligibility for the study. If there is no archival tissue a fresh biopsy will be requested from the patient. A blood sample will also be taken for future genetic analysis. Once taking part in the trial patients will need to attend their oncology unit regularly for monitoring and the delivery of treatment. Patients will undergo complete physical examination at screening, on C1D1, C1D8, C1D15, C2D1, C2D8 and day 1 of every subsequent cycle. Blood for haematology, biochemistry and clotting will be taken at each of these visits. A 12 lead ECG will be performed at screening . Disease assessment will be by CT scanning using modified RECIST criteria after 9 and 18 weeks, then every 3 months until disease progression.

DETAILED DESCRIPTION:
No further information in addition to what has been provided in the brief summary

ELIGIBILITY:
Inclusion Criteria:

* Aged >/= 16 years
* Able to provide evidence from an accredited laboratory of wt BRAF status for their melanoma, or ascertainment of wt BRAF status from a sample of melanoma provided for mutational analysis in Oxford.
* Unresectable stage 3 or 4, histologically proven cutaneous or unknown primary melanoma
* At least 1 lesion, not previously irradiated, that can be accurately measured on CT or MRI as defined by modified RECIST criteria
* ECOG performance score of 0 or 1.
* Life expectancy of at least 12 weeks.
* The patient is willing to give consent to the main study and able to comply with the protocol for the duration of the study, including scheduled follow-up visits and examinations.
* Haematological and biochemical indices within the ranges shown below. Lab Test Value required Haemoglobin (Hb) >10g/dL White Blood Count (WBC) > 3x109/L Platelet count > 100,000/μL Absolute Neutrophil count > 1.5x109/L; Serum bilirubin ≤ 1.2 x ULN AST (SGOT) or ALT ≤ 2.5 x ULN LDH ≤ 2 x ULN Creatinine clearance (Cockcroft-Gault) >50 ml/min

Exclusion Criteria:

* Any anti-cancer therapy (including radiotherapy and participation in other clinical trials) within 28 days prior to Day 1.
* Prior DNA damaging agents or cytotoxic chemotherapy for metastatic melanoma.
* Any unresolved toxicity from prior anti-cancer therapy that is greater than CTCAE grade 2.
* Pregnancy or breastfeeding women. Female patients must have a negative urinary or serum pregnancy test or have evidence of post-menopausal status (defined as absence of menstruation for > 12 months, bilateral oophrectomy or hysterectomy).
* Grade ≥2 peripheral neuropathy at study entry.
* Patients of reproductive potential who are not willing to use adequate contraceptive measures for the duration of the study (both male and female patients)
* Known severe hypersensitivity reactions to docetaxel or other drugs formulated in polysorbate 80
* Ocular or mucosal malignant melanoma
* Another active malignancy within the past five years.
* Evidence of brain metastases, unless surgically resected/stereotactic radiosurgery treated brain metastasis with no evidence of relapse on cerebral MRI, or treated brain metastasis and stable off treatment, including steroids, for 3 months.
* Clinically significant and uncontrolled major medical condition(s): such as active infection, bleeding diathesis.
* Patients who are known to be serologically positive for Hepatitis B, Hepatitis C or HIV.
* Cardiac conditions, including uncontrolled hypertension (BP>160/100 despite treatment), heart failure NYHA class 2 or above, prior or current cardiomyopathy, myocardial infarction within 6 months or angina requiring nitrate therapy more than once a week.
* Previous treatment with EGFR, ras, raf or MEK inhibitors.
* Inability to swallow capsules, refractory nausea and vomiting, chronic gastrointestinal diseases (eg, inflammatory bowel disease) or significant bowel resection that would preclude adequate absorption.
* Taking medication that significantly induces or inhibits CYP3A4.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Middleton, Principal Investigator — University of Oxford
Locations (1):
- Churchill Hospital, Oxford, Oxfordshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of 83 participants from 16 centres (hospitals) took place between October 2010 and May 2012. Participants attended clinic visits according to the protocol.
Period: Overall Study
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Started | 41 | 42
Completed (Numbers completed here are those who started treatment i.e. only excludes those who received no allocated intervention. Treatment duration is flexible, there is not mark for treatment completion, patients can keep receiving cycles of treatment up to 6 cycles.) | 38 | 41
Not Completed | 3 | 1
Not completed — Randomised, later found to be ineligible and did not start treatment | 1 | 1
Not completed — Randomised and found to be too unwell to start treatment | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomised patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (12.0) | 59.2 (13.3) | 59.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 25
  Male | 31 | 27 | 58
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 41 | 42 | 83
Stage [Count of Participants; unit: Participants] — M0 = No distant metastases M1a = Distant skin, subcutaneous, or nodal metastases (normal serum LDH) M1b = Lung metastases (normal serum LDH) M1c = All other visceral metastases (normal serum LDH); Any distant metastasis (elevated LDH)
  Participants
    M1c | 33 | 32 | 65
    M0 or M1a or M1b | 8 | 10 | 18
ECOG Performance Score [Count of Participants; unit: Participants] — 0 = Fully active, able to carry out all on all pre-disease performance without restriction. 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light housework, office work. 2 = Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours. 3 = Capable of only limited self-care. Confined to bed or chair more than 50% of waking hours. 4 = Completely disabled. Cannot carry out any self-care. Totally confined to bed or chair.
  Participants
    0 | 28 | 34 | 62
    1 | 13 | 8 | 21
Smoking status [Count of Participants; unit: Participants]
  Yes | 4 | 3 | 7
  No, but smoked in the past | 22 | 27 | 49
  Never smoked | 15 | 12 | 27
Physical examination [Count of Participants; unit: Participants] — n =Freq of pts with abnormal results. Physical examination undertaken in line with established clinical practice, adhering specifically to the standards required as part of UK medical training. Outputs from such an examination are diverse and not usually, in and of themselves, definitive. Rather they point to potential system specific abnormalities evaluated further so as to identify the issue, its severity and relationship to IMPs. Population: Not all patients were evaluated for each abnormality
  Participants
    General appearance: number analyzed (Participants) | 39 | 42 | 81
    General appearance | 0 | 1 | 1
    Skin | 21 | 13 | 34
    HEENT: number analyzed (Participants) | 36 | 40 | 76
    HEENT | 1 | 4 | 5
    Chest: number analyzed (Participants) | 39 | 42 | 81
    Chest | 4 | 5 | 9
    Cardiovascular: number analyzed (Participants) | 39 | 42 | 81
    Cardiovascular | 0 | 0 | 0
    Abdomen: number analyzed (Participants) | 39 | 42 | 81
    Abdomen | 5 | 2 | 7
    Lymph nodes: number analyzed (Participants) | 37 | 41 | 78
    Lymph nodes | 7 | 8 | 15
    Extremities/back: number analyzed (Participants) | 39 | 41 | 80
    Extremities/back | 7 | 7 | 14
    Musculoskeletal: number analyzed (Participants) | 34 | 40 | 74
    Musculoskeletal | 2 | 4 | 6
    Neurological: number analyzed (Participants) | 34 | 40 | 74
    Neurological | 1 | 2 | 3
    Other body system: number analyzed (Participants) | 37 | 40 | 77
    Other body system | 2 | 4 | 6
Vital Signs: temperature [Median (Full Range); unit: degrees C] — Population: Totals are patients with available data
  degrees C
    number analyzed (Participants) | 40 | 40 | 80
    (all) | 36.2 [35.2 to 37.3] | 36.5 [35 to 37.4] | 36.4 [35 to 37.4]
Height [Mean (Standard Deviation); unit: meters] | 1.74 (0.1) | 1.70 (0.1) | 1.72 (0.1)
Weight [Mean (Standard Deviation); unit: kg] | 88.4 (19.0) | 83.0 (19.5) | 85.7 (19.3)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 2.022 (0.232) | 1.939 (0.260) | 1.980 (0.249)
Biochemistry [Median (Full Range); unit: U/L] — Population: Numbers analysed are available data
  U/L
    ALT: number analyzed (Participants) | 41 | 41 | 82
    ALT | 26 [7 to 93] | 22 [6 to 54] | 24 [6 to 93]
    AST: number analyzed (Participants) | 37 | 38 | 75
    AST | 24 [12 to 104] | 22 [14 to 58] | 23 [12 to 104]
LDH [Count of Participants; unit: Participants]
  Above Upper limit normal | 20 | 27 | 47
  Below Upper limit normal | 21 | 15 | 36
Haematology [Median (Full Range); unit: cells x 10^9/L] — Population: Numbers analysed are those with available data
  cells x 10^9/L
    White cell count: number analyzed (Participants) | 41 | 41 | 82
    White cell count | 8 [4 to 15] | 7 [5 to 13] | 8 [4 to 19]
    Neutrophils: number analyzed (Participants) | 41 | 41 | 82
    Neutrophils | 5 [2 to 11] | 5 [2 to 11] | 5 [2 to 17]
    Platelets: number analyzed (Participants) | 41 | 41 | 82
    Platelets | 259 [147 to 681] | 255 [177 to 754] | 259 [147 to 754]
Abnormal ECG [Count of Participants; unit: Participants] — N=abnormal electrocardiogram Population: Number Analyzed represents the number of participants evaluated for this Baseline Measure
  Participants
    number analyzed (Participants) | 41 | 41 | 82
    (all) | 4 | 4 | 8
Abnormal Urinalysis [Count of Participants; unit: Participants] — N= abnormal urinalysis Population: Number Analyzed represents the number of participants evaluated for this Baseline Measure
  Participants
    number analyzed (Participants) | 39 | 38 | 77
    (all) | 9 | 8 | 17
Conmeds [Count of Participants; unit: Participants] — Number of patients reporting taking con meds at baseline
  Participants | 35 | 33 | 68
Target lesion Sum LD [Median (Full Range); unit: mm] — Site, location & longest diameter (LD) for each of up to 10 measurable Target Lesions (TL) measured. At baseline the sum of the LD for all TL is reported as baseline sum LD. At follow-up visits the sum of the LD for all TL is reported as follow-up LD.
  mm | 98 [16 to 243] | 56 [11 to 450] | 71 [11 to 450]
Vital Signs: Pulse rate [Median (Full Range); unit: Beats per minutes] — Population: Totals are patients with available data
  Beats per minutes
    number analyzed (Participants) | 41 | 41 | 82
    (all) | 70 [56 to 100] | 72 [42 to 120] | 71.5 [42 to 120]
Vital Signs: Systolic blood pressure [Median (Full Range); unit: mmHg] — Population: Totals are patients with available data
  mmHg
    number analyzed (Participants) | 41 | 41 | 82
    (all) | 137 [97 to 192] | 136 [113 to 175] | 137 [97 to 192]
Diastolic BP [Median (Full Range); unit: mmHg] — Population: Totals are patients with available data
  mmHg
    number analyzed (Participants) | 41 | 41 | 82
    (all) | 85 [56 to 115] | 82 [68 to 95] | 83.5 [56 to 115]
Biochemistry: Bilirubin [Median (Full Range); unit: µmol/L] — Population: Numbers analysed are available data
  µmol/L
    number analyzed (Participants) | 41 | 41 | 82
    (all) | 10 [4 to 21] | 8 [2 to 18] | 9 [2 to 21]
Biochemistry: Creatine clearance [Median (Full Range); unit: ml/min] — Population: Numbers analysed are available data
  ml/min
    number analyzed (Participants) | 40 | 41 | 81
    (all) | 111 [54 to 233] | 94 [39 to 194] | 98 [39 to 233]
Haematology: Haemoglobin [Median (Full Range); unit: g/dL] — Population: Numbers analysed are those with available data
  g/dL
    number analyzed (Participants) | 41 | 41 | 82
    (all) | 14 [10 to 16] | 14 [10 to 17] | 14 [10 to 17]

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: This is defined as time from date of randomisation to the first of date of progression (using CT scan, x-ray, MRI scan and clinical examination) using modified RECIST (v1.1) criteria or date of death (events). For patients without an event, the time from date of randomisation to date last known alive will be the censored PFS time.
Time Frame: From randomisation date to date of PFS event, if they did not have an event by the end of trial datalock (01Oct2012), an average of 9.3 months.
Population: The primary analysis was intention to treat and involved all patients who were randomly assigned.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 41 | 42
months | 4.23 [3.63 to 6.90] | 3.93 [2.07 to 4.16]
Statistical Analysis 1: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; Test type: Superiority; p = 0.130, Regression, Cox — p value < 0.1 one-sided considered to be significant; Hazard Ratio (HR) = 0.753, 90% CI 2-sided [0.498 to 1.138] — HR is Adjusted for M status, performance status
Statistical Analysis 2: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; This is a sensitivity analysis of the primary outcome. This includes all 83 patients but the analysis additionally adjusted for LDH, target lesion sum and time interval between randomisation and baseline CT scan as well as mstatus, performance status; Test type: Superiority; p = 0.113, Regression, Cox; Hazard Ratio (HR) = 0.723, 90% CI 2-sided [0.465 to 1.123] — This includes all 83 patients but the analysis additionally adjusted for LDH, target lesion sum and time interval between randomisation and baseline CT scan as well as mstatus, performance status
Statistical Analysis 3: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; This is a sensitivity analysis, including all 83 randomised patients. Patients are assessed periodically for the response (progression), the time when the event occurred is not directly observed but is known to take place within some time interval. Progression is known only to have occurred at some time between visits, the exact time is not known. We carried out interval censored analysis to demonstrate if allowing for interval censoring gives a different interpretation of the primary outcome; Test type: Superiority; p = 0.3016, Generalised log-rank — This analysis assesses if allowing for interval censoring is consistent with the primary outcome results; Generalised log-rank taking into account interval censoring, analysed using SAS package version 9.2. Method by Zhao and Sun, 2004
Statistical Analysis 4: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; Sensitivity analysis adjusting for centre. All 83 randomised patients were included in analysis. Centres were the three biggest recruiters and all other 13 centres are combined; Test type: Superiority; p = 0.305, Regression, Cox; Hazard Ratio (HR) = 1.348, 90% CI 2-sided [0.602 to 3.016] — Adjusted for centre

2. Secondary Outcome: Progression Free Survival Rate at 6 Months
Description: PFS at 6 months is defined as the percentage progression free survival at 6 months from the PFS Kaplan Meier graph. This would allow all patients randomised to be included. progression was diagnosed using CT scan, x-ray, MRI scan and clinical examination using modified RECIST(v1.1) criteria.
Time Frame: as for outcome 1
Population: Intention to treat i.e. all randomised patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 41 | 42
percentage of participants | 40 [27 to 53] | 26 [15 to 38]
Statistical Analysis 1: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; Test type: Superiority; p = 0.187, Log Rank; Mean Difference (Final Values) = 14, 90% CI 2-sided [-3.4 to 31.4] — This is the estimated difference in PFS rate i.e. % difference between arms

3. Secondary Outcome: Overall Survival
Description: This is defined as the time from randomisation to death (event) or time from randomisation to date last known alive (censored time).
Time Frame: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 41 | 42
months | 9.5 [8.467 to 12.9] | 11.367 [7.467 to 18]
Statistical Analysis 1: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; Test type: Superiority; p = 0.169, Regression, Cox; p value < 0.1 one-sided considered to be significant; Hazard Ratio (HR) = 1.373, 90% CI 2-sided [0.797 to 2.369]

4. Secondary Outcome: Objective Response Rate
Description: Objective response rate calculated as number of patients with Complete Response (CR) or Partial response (PR) over all patients randomised. The numerator of the objective response rate is the number of patients achieving a CR or PR. The denominator is all patients randomised. RECIST(v1.1) criteria was used for assessment.
Time Frame: as for outcome 1
Population: intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 41 | 42
Participants
  Complete response | 1 | 0
  Partial response | 12 | 6
  Stable disease | 14 | 15
  Progressive disease | 5 | 19
  Not applicable | 9 | 2
Statistical Analysis 1: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; Objective response rate calculated as number of patients with CR or PR over all patients randomised; Test type: Superiority; p = 0.059, Chi-squared

5. Secondary Outcome: Overall Survival Results - Post Final Analysis
Description: OS analysis was carried out at the final analysis time point on data taken on 01Oct2012. Another data extraction was taken on 05Mar2013 in order to carry out posthoc analyses, OS was analysed again on this data.
  OS is time from randomisation to death (event) or time from randomisation to date last known alive (censored time).
Time Frame: as for outcome 1
Population: Intention to treat
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 41 | 42
months | 9.5 [8.47 to 12.53] | 11.37 [8.67 to 16.03]
Statistical Analysis 1: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; Analysis adjusted for with Mstatus and Performance Score; Test type: Superiority; p = 0.318, Regression, Cox; Hazard Ratio (HR) = 1.15, 90% CI 2-sided [0.71 to 1.84]

6. Secondary Outcome: Vital Signs - Temperature
Description: Vital signs - temperature.
Time Frame: From randomisation date to date of PFS event, if they did not have an event by the end of trial datalock (01Oct2012), an average of 9.3 months. Reported value for each arm is median value across all time-points for all patients in that arm.
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: Degree celsius
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 361 | 371
Degree celsius | 36.2 [35.9 to 36.6] | 36.3 [35.9 to 36.7]

7. Secondary Outcome: Vital Signs - Pulse Rate
Description: Vital signs - pulse rate.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: Beats per minute
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 374 | 377
Beats per minute | 78 [69 to 88] | 84 [72 to 96]

8. Secondary Outcome: Vital Signs - Systolic Blood Pressure
Description: Vital signs - systolic blood pressure.
Time Frame: as for outcome 6
Population: Whole study
Measure: Median (Inter-Quartile Range); unit: Mg mercury
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 375 | 379
Mg mercury | 131 [121 to 144] | 130 [120 to 140]

9. Secondary Outcome: Vital Signs - Diastolic Blood Pressure
Description: Vital signs - diastolic blood pressure.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: Mg mercury
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 375 | 378
Mg mercury | 82 [73 to 90] | 79 [71 to 85]

10. Secondary Outcome: Weight
Description: Weight.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: Kg
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 39 | 40
Number analyzed (Data points) | 320 | 317
Kg | 90.425 [80.95 to 99.1] | 83.45 [68.2 to 96.7]

11. Secondary Outcome: Haematology - Haemoglobin
Description: Haematology - haemoglobin.
Time Frame: as for outcome 6
Population: Whole study
Measure: Median (Inter-Quartile Range); unit: grams per litre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 385 | 400
grams per litre | 12.5 [11.6 to 13.6] | 12.9 [11.7 to 13.9]

12. Secondary Outcome: Haematology - White Cell Count
Description: Haematology - white cell count.
Time Frame: From randomisation date to date of PFS event, if they did not have an event by the end of trial datalock (01Oct2012), an average of 9.3 months. Reported values for each arm are median values across all time-points for all patients in that arm.
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: 10^9 cells litre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 386 | 400
10^9 cells litre | 7.75 [5.1 to 11.2] | 8.405 [4.84 to 13.295]

13. Secondary Outcome: Haematology - Neutrophils
Description: Haematology - neutrophils.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: 10^9 cells litre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 385 | 400
10^9 cells litre | 5.4 [2.64 to 8.82] | 5.7 [2.85 to 11.46]

14. Secondary Outcome: Haematology - Platelets
Description: Haematology - platelets.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: 10^9 cells litre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 385 | 400
10^9 cells litre | 267 [223 to 324] | 290.5 [229.5 to 363]

15. Secondary Outcome: Biochemistry - Phosphate
Description: Biochemistry - phosphate.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: mmol per litre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 40
Number analyzed (Data points) | 350 | 346
mmol per litre | 1.245 [1.08 to 1.43] | 1 [0.86 to 1.16]

16. Secondary Outcome: Biochemistry - Calcium
Description: Biochemistry - calcium.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: mmol per litre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 373 | 384
mmol per litre | 2.28 [2.2 to 2.36] | 2.34 [2.26 to 2.43]

17. Secondary Outcome: Biochemistry - Sodium
Description: Biochemistry - sodium.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: mmol per litre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 383 | 396
mmol per litre | 139 [137 to 141] | 139 [137 to 140]

18. Secondary Outcome: Biochemistry - Potassium
Description: Biochemistry - potassium.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: mmol per litre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 379 | 389
mmol per litre | 4.3 [4 to 4.54] | 4.3 [4 to 4.6]

19. Secondary Outcome: Biochemistry - Urea
Description: Biochemistry - urea.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: mmol per litre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 383 | 393
mmol per litre | 5.7 [4.7 to 6.6] | 5.2 [4.1 to 6.4]

20. Secondary Outcome: Biochemistry - Bilirubin
Description: Biochemistry - bilirubin.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: umol per litre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 380 | 391
umol per litre | 7 [5 to 10] | 7 [5 to 10]

21. Secondary Outcome: Biochemistry - Alkaline Phosphatase
Description: Biochemistry - alkaline phosphatase.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: IU per litre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 383 | 394
IU per litre | 93 [72 to 147] | 85 [64 to 153]

22. Secondary Outcome: Biochemistry - ALT
Description: Biochemistry - ALT.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: IU per litre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 380 | 390
IU per litre | 32 [23 to 47] | 21 [16 to 31]

23. Secondary Outcome: Biochemistry - AST
Description: Biochemistry - AST.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: IU per litre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 38 | 39
Number analyzed (Data points) | 308 | 351
IU per litre | 32 [25 to 41] | 20 [17 to 26]

24. Secondary Outcome: Biochemistry - Albumin
Description: Biochemistry - albumin.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: grams per litre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 383 | 394
grams per litre | 37 [34 to 41] | 40 [37 to 43]

25. Secondary Outcome: Biochemistry - GGT
Description: Biochemistry - GGT.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: grams per litre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 354 | 357
grams per litre | 41 [26 to 73] | 30 [20 to 52]

26. Secondary Outcome: Biochemistry - Total Protein
Description: Biochemistry - total protein.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: grams per litre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 377 | 378
grams per litre | 66 [62 to 71] | 67 [63 to 71]

27. Secondary Outcome: Biochemistry - LDH
Description: Biochemistry - LDH.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: Units per litre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 339 | 326
Units per litre | 305 [243 to 491] | 386.5 [233 to 499]

28. Secondary Outcome: Biochemistry - Creatinine
Description: Biochemistry - creatinine.
Time Frame: as for outcome 6
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: milligrams per decalitre
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 39 | 41
Number analyzed (Data points) | 334 | 346
milligrams per decalitre | 113.6 [94 to 139.26] | 98.3 [83.5 to 119.18]

29. Secondary Outcome: Physical Assessment - General Appearance
Description: Physical assessment - general appearance.
Time Frame: From randomisation date to date of PFS event, if they did not have an event by the end of trial datalock (01Oct2012), an average of 9.3 months. Reported values for each arm are total counts across all time-points for all patients in that arm.
Population: Intention to treat
Measure: Count of Units; unit: Data points
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 34 | 36
Number analyzed (Data points) | 234 | 198
Data points
  Normal | 181 | 162
  Abnormal | 35 | 24
  Not evaluated | 18 | 12

30. Secondary Outcome: Physical Exam - Skin
Description: Physical exam - skin.
Time Frame: as for outcome 29
Population: Intention to treat
Measure: Count of Units; unit: Data points
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 34 | 36
Number analyzed (Data points) | 234 | 197
Data points
  Normal | 56 | 86
  Abnormal | 155 | 99
  Not evaluated | 23 | 12

31. Secondary Outcome: Physical Exam - Head and Neck
Description: Physical exam - head and neck.
Time Frame: as for outcome 29
Population: Intention to treat
Measure: Count of Units; unit: Data points
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 34 | 36
Number analyzed (Data points) | 234 | 197
Data points
  Normal | 139 | 146
  Abnormal | 61 | 23
  Not evaluated | 34 | 28

32. Secondary Outcome: Physical Exam - Chest
Description: Physical exam - chest.
Time Frame: as for outcome 29
Population: Intention to treat
Measure: Count of Units; unit: Data points
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 34 | 36
Number analyzed (Data points) | 234 | 197
Data points
  Normal | 187 | 170
  Abnormal | 29 | 16
  Not evaluated | 18 | 11

33. Secondary Outcome: Physical Exam - Cardiovascular
Description: Physical exam - cardiovascular.
Time Frame: as for outcome 29
Population: Intention to treat
Measure: Count of Units; unit: Data points
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 34 | 36
Number analyzed (Data points) | 234 | 197
Data points
  Normal | 204 | 180
  Abnormal | 7 | 6
  Not evaluated | 23 | 11

34. Secondary Outcome: Physical Exam - Abdomen
Description: Physical exam - abdomen.
Time Frame: as for outcome 29
Population: Intention to treat
Measure: Count of Units; unit: Data points
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 34 | 36
Number analyzed (Data points) | 234 | 197
Data points
  Normal | 205 | 163
  Abnormal | 5 | 24
  Not evaluated | 24 | 10

35. Secondary Outcome: Physical Exam - Lymph Nodes
Description: Physical exam - lymph nodes.
Time Frame: as for outcome 29
Population: Intention to treat
Measure: Count of Units; unit: Data points
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 34 | 36
Number analyzed (Data points) | 234 | 197
Data points
  Normal | 162 | 148
  Abnormal | 19 | 27
  Not evaluated | 53 | 22

36. Secondary Outcome: Physical Exam - Extremities
Description: Physical exam - extremities.
Time Frame: as for outcome 29
Population: Intention to treat
Measure: Count of Units; unit: Data points
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 34 | 36
Number analyzed (Data points) | 234 | 197
Data points
  Normal | 114 | 139
  Abnormal | 83 | 37
  Not evaluated | 37 | 21

37. Secondary Outcome: Physical Exam - Musculoskeletal
Description: Physical exam - musculoskeletal.
Time Frame: as for outcome 29
Population: Intention to treat
Measure: Count of Units; unit: Data points
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 34 | 36
Number analyzed (Data points) | 234 | 197
Data points
  Normal | 156 | 149
  Abnormal | 19 | 13
  Not evaluated | 59 | 35

38. Secondary Outcome: Physical Exam - Neurological
Description: Physical exam - neurological.
Time Frame: as for outcome 29
Population: Intention to treat
Measure: Count of Units; unit: Data points
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 34 | 36
Number analyzed (Data points) | 234 | 197
Data points
  Normal | 149 | 129
  Abnormal | 7 | 19
  Not evaluated | 78 | 49

39. Secondary Outcome: Physical Exam - Other
Description: Physical exam - other.
Time Frame: as for outcome 29
Population: Intention to treat
Measure: Count of Units; unit: Data points
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 19 | 13
Number analyzed (Data points) | 52 | 47
Data points
  Normal | 4 | 4
  Abnormal | 40 | 31
  Not evaluated | 8 | 12

40. Secondary Outcome: ECG - Pre-dose
Description: ECG - pre-dose.
Time Frame: as for outcome 29
Population: Intention to treat
Measure: Count of Units; unit: Data points
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 40 | 41
Number analyzed (Data points) | 67 | 122
Data points
  Normal | 39 | 39
  Abnormal | 5 | 6
  Not evalauated | 23 | 77

41. Secondary Outcome: ECG - Post-dose
Description: ECG - post-dose.
Time Frame: as for outcome 29
Population: Intention to treat
Measure: Count of Units; unit: Data points
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 39 | 41
Number analyzed (Data points) | 68 | 127
Data points
  Normal | 32 | 34
  Abnormal | 5 | 6
  Not evaluated | 31 | 87

42. Secondary Outcome: Urinalysis
Description: Urinalysis.
Time Frame: as for outcome 29
Population: Intention to treat
Measure: Count of Units; unit: Data points
Units Other Than Participants: Data points
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 39 | 41
Number analyzed (Data points) | 372 | 365
Data points
  Normal | 205 | 229
  Abnormal | 130 | 117
  Not evaluated | 37 | 19

43. Other Pre Specified Outcome: Progression Free Survival: Sensitivity Analysis 1
Description: Same as for primary analysis. This is defined as time from date of randomisation to the first of date of progression (using CT scan, x-ray, MRI scan and clinical examination) using modified RECIST v1.1 criteria or date of death (events). For patients without an event, the time from date of randomisation to date last known alive will be the censored PFS time.
Time Frame: as for outcome 1
Population: This is a sensitivity analysis of the primary outcome and includes randomised patients that had CT scans as per protocol.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 28 | 33
months | 4.1 [2.1 to 4.233] | 3.333 [2.067 to 4.167]
Statistical Analysis 1: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; This is a sensitivity analysis of the primary outcome; Test type: Superiority; p = 0.468, Regression, Cox; Hazard Ratio (HR) = 1.022, 90% CI 2-sided [0.649 to 1.612] — Analysis Adjusted for M status, performance status

44. Other Pre Specified Outcome: Progression Free Survival- Per Protocol Analysis
Description: Same as for primary analysis. This is defined as time from date of randomisation to the first of date of progression (using CT scan, x-ray, MRI scan and clinical examination) using modified RECIST v1.1. criteria or date of death (events). For patients without an event, the time from date of randomisation to date last known alive will be the censored PFS time.
Time Frame: as for outcome 1
Population: Per-protocol population, this is the primary analysis population excluding four patients who did not start treatment and two patients who were later found to be ineligible.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 37 | 40
months | 4.3 [4.1 to 7.033] | 4.067 [2.1 to 4.2]
Statistical Analysis 1: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; This is the per-protocol analysis of the primary outcome; Test type: Superiority; p = 0.106, Regression, Cox; Hazard Ratio (HR) = 0.721, 90% CI 2-sided [0.468 to 1.109] — Analysis was adjusted for mstatus, performance status

45. Post Hoc Outcome: Progression Free Survival: in Patients With NRAS Data
Description: Outcome is time from randomisation to progression or death in subset of patients with NRAS mutational data available and in the per-protocol population.
  progression was diagnosed using CT scan, x-ray, MRI scan and clinical examination using modified RECIST(v1.1) criteria.
  NRAS mutational analysis (wild type or mutated) for all patients was derived from archival melanoma tumour tissue samples.
Time Frame: as for outcome 1
Population: per protocol population and only those with NRAS status
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 29 | 31
months | 4.4 [3.4 to 7.13] | 4.1 [2.07 to 4.2]
Statistical Analysis 1: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; Model with interaction term between NRAS status and treatment group and stratification variables; Test type: Superiority; p = 0.824, Regression, Cox — p-value is for the interaction term; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.25 to 1.53] — HRs (95% CI) between treatment groups are given for Wild type and NRAS mutated separately. The above HR is for WT

46. Post Hoc Outcome: Overall Survival in Patients With NRAS Data
Description: Outcome is time from randomisation to death in subset of patients with NRAS mutational data available and in the per-protocol population.
  NRAS mutational analysis (wild type or mutated) for all patients was derived from archival melanoma tumour tissue samples.
Time Frame: as for outcome 1
Population: Per protocol population and only those with NRAS data
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 29 | 31
months | 12.07 [8.47 to 12.9] | 11.9 [9.3 to 18]
Statistical Analysis 1: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; Test type: Superiority; p = 0.072, Regression, Cox — p-value is for interaction term; Model includes interaction term between NRAS status and treatment group and stratification variables; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.16 to 1.60] — HRs for treatment effect (AZD6244 vs Placebo ) are estimated for NRAS WT and NRAS mutated patients separately. Hazard ratios (95%CI) given above are for NRAS WT patients
Statistical Analysis 2: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.97, 95% CI 2-sided [0.73 to 5.33] — HR for NRAS mutated patients

47. Post Hoc Outcome: Objective Response Rate in Patients With WT NRAS
Description: Best overall response as reported for evaluable/measurable scans including target, non-target and new lesions. Response assessed using RECIST(v1.1) criteria.
  Data from Mar2013 which was post final data lock
Time Frame: as for outcome 1
Population: Per protocol population and only those with NRAS status- wild type
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 9 | 14
Participants
  Complete response | 0 | 0
  Partial response | 2 | 2
  Stable disease | 4 | 4
  Progressive disease | 3 | 8
  Not applicable | 0 | 0

48. Post Hoc Outcome: Overall Survival Results - Post Final Analysis- Per-protocol
Description: as for outcome 5
Time Frame: as for outcome 1
Population: Per protocol population.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 37 | 40
months | 10.9 [8.53 to 12.53] | 11.77 [8.67 to 16.03]
Statistical Analysis 1: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; Test type: Superiority — Adjusted for with Mstatus and Performance Score; p = 0.348, Regression, Cox; Hazard Ratio (HR) = 1.12, 90% CI 2-sided [0.68 to 1.87]

49. Post Hoc Outcome: Progression Free Survival: in Patients With NRAS Data- Sensitivity
Description: Outcome is time from randomisation to progression or death in subset of patients with NRAS mutational data available and in the per-protocol population and excluding patients found to have BRAF mutation on retesting (the inclusion criteria for the trial is those with wildtype BRAF).
  progression was diagnosed using CT scan, x-ray, MRI scan and clinical examination using modified RECIST(v1.1) criteria.
  NRAS mutational analysis (wild type or mutated) for all patients was derived from archival melanoma tumour tissue samples.
Time Frame: as for outcome 1
Population: per-protocol population and only patients with NRAS mutational data and excluding patients found to have BRAF mutation on retesting
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 28 | 30
months | 4.4 [3.4 to 7.27] | 4.1 [2.07 to 4.27]
Statistical Analysis 1: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; Test type: Superiority; p = 0.797, Regression, Cox — p-value is for interaction term; Model includes interaction term between NRAS status and treatment group and stratification variables; Hazard Ratio (HR) = 0.61, 90% CI 2-sided [0.24 to 1.58] — [estimate comment as in outcome 46, analysis 1]
Statistical Analysis 2: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.350 to 1.45] — HR for NRAS mutated patients

50. Post Hoc Outcome: Overall Survival in Patients With NRAS Data- Sensitivity
Description: Outcome is time from randomisation to death in subset of patients with NRAS mutational data available and in the per-protocol population and excluding patients found to have BRAF mutation on retesting (the inclusion criteria for the trial is those with wildtype BRAF).
  NRAS mutational analysis (wild type or mutated) for all patients was derived from archival melanoma tumour tissue samples.
Time Frame: as for outcome 1
Population: Per-protocol population, including only patients with NRAS data and excluding patients found to have BRAF mutation on retesting
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 28 | 30
months | 12.07 [8.47 to 12.9] | 11.9 [10.43 to 18]
Statistical Analysis 1: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; Test type: Superiority; p = 0.120, Regression, Cox — Model includes interaction term between NRAS status and treatment group and stratification variables. p-value is for interaction term; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.18 to 1.97] — [estimate comment as in outcome 46, analysis 1]
Statistical Analysis 2: Comparison: Docetaxel and AZD6244 vs Docetaxel and Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.99, 95% CI 2-sided [0.73 to 5.38] — HR for NRAS mutated patients

51. Post Hoc Outcome: Objective Response Rate in Patients With Mutated NRAS
Description: as for outcome 47
Time Frame: as for outcome 1
Population: Per protocol population and only those with NRAS status=mutated
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
Number analyzed (Participants) | 20 | 17
Participants
  Complete response | 1 | 0
  Partial response | 6 | 2
  Stable disease | 7 | 9
  Progressive disease | 2 | 6
  Not applicable | 4 | 0

ADVERSE EVENTS:
Time Frame: 170 days
Description: Adverse event monitoring starts from the time the patient receives any of the research procedures until 30 days post treatment (treatment was 6 3-week cycles, 126 days) and the first trial research procedure was up to 14 days prior to starting treatment. Total safety assessment time frame was a maximum of 170 days and minimum of 157 days, dependent on when the patient had their first research procedure prior to starting treatment (1-14 days).
Arm/Group | Docetaxel and AZD6244 | Docetaxel and Placebo
All-Cause Mortality (participants affected / at risk) | 26/41 | 28/42
Serious Adverse Events (participants affected / at risk) | 29/41 | 20/42
Other Adverse Events (participants affected / at risk) | 35/41 | 40/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Docetaxel and AZD6244 (N=41) | Docetaxel and Placebo (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 20 (25) | 13 (16)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Retinal Vascular Disorder (Eye disorders) | 1/1 (1) | 0/0 (0) — Retinal Vascular Disorder
Gastric Haemorrhage (Gastrointestinal disorders) | 2/2 (2) | 0 (0) — Gastric Haemorrhage
Vomiting (Gastrointestinal disorders) | 1 (1) | 1/1 (1) — Vomiting
Diarrhoea (Gastrointestinal disorders) | 2/2 (2) | 1 (1) — Diarrhoea
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Abdominal Pain
Fever (General disorders) | 5 (6) | 2 (2) — Fever
Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0) — Allergic Reaction
Other - Source Unknown (Infections and infestations) | 0 (0) | 1 (1) — Other - Source Unknown
Enterocolitis Infectious (Infections and infestations) | 0 (0) | 1 (1) — Enterocolitis Infectious
Skin Infection (Infections and infestations) | 2 (2) | 0 (0) — Skin Infection
Lung Infection (Infections and infestations) | 1 (1) | 2 (2) — Lung Infection
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0) — Upper Respiratory Infection
Sepsis (Infections and infestations) | 2 (2) | 0 (0) — Sepsis
Neutrophil Count Decreased (Investigations) | 1 (1) | 0 (0) — Neutrophil Count Decreased
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Arthralgia
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Muscle Weakness Lower Limb
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) — Presyncope
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1/1 (1) | 1 (1) — Dyspnea
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel and AZD6244 (N=41) | Docetaxel and Placebo (N=42)
Anaemia (Blood and lymphatic system disorders) | 2 (6) | 4 (5)
Febrile Neutropenia (Blood and lymphatic system disorders) | 8 (11) | 5 (6) — Febrile Neutropenia
Blurred Vision (Eye disorders) | 4 (5) | 1 (1) — Blurred Vision
Dry Eye (Eye disorders) | 2 (3) | 1 (1) — Dry Eye
Floaters (Eye disorders) | 1 (1) | 0 (0) — Floaters
Watering Eyes (Eye disorders) | 5 (7) | 5 (5) — Watering Eyes
Nausea (Gastrointestinal disorders) | 19 (30) | 15 (18) — Nausea
Constipation (Gastrointestinal disorders) | 11 (13) | 11 (15) — Constipation
Flatulence (Gastrointestinal disorders) | 1 (3) | 1 (2) — Flatulence
Dyspepsia (Gastrointestinal disorders) | 5 (8) | 10 (13) — Dyspepsia
Diarrhoea (Gastrointestinal disorders) | 32 (81) | 20 (29) — Diarrhoea
Dry Mouth (Gastrointestinal disorders) | 6 (9) | 3 (3) — Dry Mouth
Vomiting (Gastrointestinal disorders) | 11 (15) | 8 (9) — Vomiting
Abdominal Pain (Gastrointestinal disorders) | 2 (3) | 2 (2) — Abdominal Pain
Mucositis Oral (Gastrointestinal disorders) | 20 (35) | 17 (27) — Mucositis Oral
Localized Edema (General disorders) | 15 (22) | 8 (12) — Localized Edema
Fatigue (General disorders) | 28 (58) | 32 (60) — Fatigue
Fever (General disorders) | 7 (9) | 3 (3) — Fever
Allergic Reaction (Immune system disorders) | 4 (5) | 5 (7) — Allergic Reaction
Nail Infection (Infections and infestations) | 2 (2) | 0 (0) — Nail Infection
Upper Respiratory Infection (Infections and infestations) | 4 (4) | 1 (1) — Upper Respiratory Infection
Mucosal Infection (Infections and infestations) | 2 (2) | 5 (6) — Mucosal Infection
Bronchial Infection (Infections and infestations) | 0 (0) | 4 (4) — Bronchial Infection
Wound Infection (Infections and infestations) | 2 (2) | 1 (1) — Wound Infection
Urinary Tract Infection (Infections and infestations) | 2 (2) | 1 (1) — Urinary Tract Infection
Other Infection (Infections and infestations) | 3 (6) | 1 (1) — Other Infection
Skin Infection (Infections and infestations) | 5 (7) | 3 (4) — Skin Infection
Neutrophil Count Decreased (Investigations) | 4 (6) | 13 (15) — Neutrophil Count Decreased
Platelet Count Decreased (Investigations) | 0 (0) | 1 (3) — Platelet Count Decreased
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Hypoalbuminemia
Anorexia (Metabolism and nutrition disorders) | 9 (12) | 8 (11) — Anorexia
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7) | 10 (13) — Arthralgia
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 8 (11) — Myalgia
Pain - Other (Musculoskeletal and connective tissue disorders) | 17 (43) | 11 (18) — Pain - Other
Peripheral Sensory Neuropathy (Nervous system disorders) | 9 (11) | 13 (16) — Peripheral Sensory Neuropathy
Dizziness (Nervous system disorders) | 5 (11) | 4 (4) — Dizziness
Dysgeusia (Nervous system disorders) | 14 (19) | 13 (18) — Dysgeusia
Headache (Nervous system disorders) | 3 (3) | 3 (4) — Headache
Depression (Psychiatric disorders) | 6 (8) | 0 (0) — Depression
Insomnia (Psychiatric disorders) | 1 (2) | 4 (6) — Insomnia
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) — Dyspnea
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 4 (7) — Epistaxis
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (5) — Cough
Other Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Other Rash
Nail Ridging (Skin and subcutaneous tissue disorders) | 7 (8) | 9 (12) — Nail Ridging
Rash Acneiform (Skin and subcutaneous tissue disorders) | 29 (54) | 20 (26) — Rash Acneiform
Dry Skin (Skin and subcutaneous tissue disorders) | 6 (8) | 1 (1) — Dry Skin
Alopecia (Skin and subcutaneous tissue disorders) | 19 (20) | 20 (21) — Alopecia
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1) — Palmar-Plantar Erythrodysesthesia Syndrome
Periorbital Edema (Skin and subcutaneous tissue disorders) | 6 (7) | 0 (0) — Periorbital Edema
Flushing (Vascular disorders) | 3 (3) | 6 (7) — Flushing
Thromboembolic Event (Vascular disorders) | 1 (1) | 1 (1) — Thromboembolic Event
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Blood Potassium (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Chest Discomfort (General disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 3 (3) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 2 (2)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Dandruff (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Diverticular Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Extravasation (General disorders) | 1 (1) | 0 (0)
Gamma-Glutamyltransferase (Investigations) | 1 (1) | 0 (0)
Gastrooeophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Influenza Like Illness (Infections and infestations) | 1 (1) | 1 (1)
Memory Impairment (Nervous system disorders) | 1 (2) | 0 (0)
Micturition Urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Mucosal Infection (Infections and infestations) | 2 (2) | 5 (6)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Rectal Haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 1 (2)
Scab (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin Nodule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tongue Coated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth Discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth Loss (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Vaginal Discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2014-07-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT01256359/Prot_000.pdf
  • Statistical Analysis Plan (2013-02-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT01256359/SAP_001.pdf